CLINICAL TRIAL: NCT01376817
Title: Comparative Study About the Impact of Two Oil Emulsions, One of Them Formulated With MCT, LCT, Olive Oil and Omega 3 Fatty Acids Versus Another One Formulated With MCT and LCT, Administered Intravenously on Severe Acute Pancreatitis Clinical Evolution
Brief Title: Comparative Study About the Impact of Two Oil Emulsions Administered Intravenously on Severe Acute Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Dr. Daniel Cardona Pera (principal investigator), Section of Artificial Nutrition and Intravenous Mixtures, Fharmacy Service, Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ELomega3; 2007-005611-26
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2009-02

CONDITIONS: Severe Acute Pancreatitis
Keywords: Severe acute pancreatitis; total parenteral nutrition; fat emulsions; omega 3 fatty acids
MeSH Terms: conditions — Pancreatitis; Hyperphagia | interventions — soybean oil, phospholipid emulsion; Olive Oil; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega 3 (Experimental)
  Interventions: Drug: Fat emulsion with MCT, LCT, olive oil and omega 3 fatty acids
- MCT / LCT (Active Comparator)
  Interventions: Drug: Fat emulsion with MCT and LCT

INTERVENTIONS:
Drug: Fat emulsion with MCT, LCT, olive oil and omega 3 fatty acids — 40% of non-protein calories (25-30 kcal/kg/day) of total parenteral nutrition, IV (in the vein), from day 1 to day 10
  Arms: Omega 3
Drug: Fat emulsion with MCT and LCT — 40% of non-protein calories (25-30 kcal/kg/day) of total parenteral nutrition, IV (in the vein), from day 1 to day 10
  Arms: MCT / LCT

SUMMARY:
The purpose of this study is to comparatively assess the potential antiinflammatory effects of intravenous lipid emulsions rich in omega 3 polyunsaturated fatty acids and olive oil versus intravenous lipid emulsions made exclusively with MCT and LCT on the evolution of patients with severe acute pancreatitis during the period in needing artificial nutrition support with total parenteral nutrition so unique.

DETAILED DESCRIPTION:
Information recorded in other data elements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pancreatitis: characteristic abdominal pain, serum amylase and / or lipase >= 3 times the upper limit of normal range, characteristic CT-scan
* Criteria of severity of acute pancreatitis diagnosed at <= 72 hours following admission: severity Index of Balthazar's CT-scan (with contrast) >= grade D, APACHE-II >= 8, C-reactive protein >= 150 mg/L
* Inability to initiate feeding (oral or with nutritional supplements) and / or enteral nutrition during the 5 days after the diagnosis and prediction of the indication of nil-by-mouth >= 5 days
* <= 3 mmol/L of triglycerides in the blood
* Men and women aged >= 18 years old
* Acceptance of informed consent

Exclusion Criteria:

* Known hipersensitivity to the fish, egg or soy proteins
* Lipid etiology
* > 3 mmol/L of triglycerides in the blood
* Severe hepatic impairment
* Severe renal insufficiency without dialysis or haemofiltration
* Serious disturbances of blood clotting
* Acute shock
* Infusion therapy general contraindications
* Clinical conditions of instability that must not be taken with parenteral nutrition
* Have other acute or chronic inflammatory diseases
* Status of severe immunosuppression: cytotoxic treatment in 15 days prior to inclusion and / or a disease that causes white blood cells levels <5000/mm3
* Treatment with steroids > 0.25 mg/kg/day of prednisone or equivalent doses of corticosteroids: as pre-treatment and / or during admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers | Day 10
  LTB4, TXB2, PG2, IL-6, alfa-TNF, C-reactive protein (CRP) Day 1 (before treatment), 5 and 10

SECONDARY OUTCOMES:
Evolution of the degree of severity of acute severe pancreatitis | During the first 72 hours after admission
  At hospital admission: age, BMI, organ failure. Evolution of the degree of severity of acute severe pancreatitis: severity risk factors at the hospital admission (age, BMI, organ failure), pronostic signs of severity during the first 72 hours after admission : APACHE-II, Ranson criteria, serum hematocrit, CT-scan with Balthazar index, CRP.
  Day 10: CT-scan with Balthazar index, CRP.
Complications of acute severe pancreatitis | Day 10.
  From day 1 to day 10. Complications of acute severe pancreatitis: local complications (necrosis, pseudocyst, abscess, surgery, ERCP), systemic complications (SIRS, sepsis, organ failure, other ones, mortality).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cardona Pera, Doctor, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- See also: Hospital de la Santa Creu i Sant Pau's website — http://www.santpau.cat/